CLINICAL TRIAL: NCT03802825
Title: Addressing Social Determinants of Health & Diabetes Self-Management in Vulnerable Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R34DK119853-01 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2019-01-14 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Eligibility criteria for all study participants is a diagnosis of diabetes with A1C ≥ 8.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation (Active Comparator): Participants randomized to the patient navigation only arm will be referred to a KPNW patient navigator using a standard electronic health record-based referral process. Once the participant has completed the Your Current Life Situation (YCLS) assessment with study staff, the navigator will receive the referral and follow-up with the participant to address the social and economic needs identified. The patient navigator will follow-up with the participant 2-3 times over the 6 month period by phone or in-person about progress with the referral and help address additional needs that may develop during the 6-month intervention. Participant will also receive monthly mailing of American Diabetes Association educational materials.
  Interventions: Other: Standard Patient Navigation
- Patient Navigation+Diabetes Self-Management Support (Experimental): In addition to receiving patient navigation as described, participants in this arm will also be referred to Project Access NOW by study staff using REDCap. Project Access NOW will connect participants to a community-based organization based on their preference, previous experience with an agency, geography, and capacity.
  The CHW will follow-up with the participant to conduct a home visit and follow-up on community-based referrals already placed by the KPNW patient navigator and assess for additional needs. The timing of the diabetes self-management training will be based on the needs of the participant.
  Interventions: Behavioral: Diabetes Self-Management Training

INTERVENTIONS:
Behavioral: Diabetes Self-Management Training — The Decision-making Education for Choices in Diabetes Everyday (DECIDE) program is a nine-module, literacy adapted diabetes and cardiovascular disease education and problem-solving training program. Participants are taught the five steps of problem solving with each module going in depth on a single step: 1) identify the problem; 2) brainstorm possible strategies for problem resolution; 3) select the most appropriate strategy; 4) apply the strategy; 5) evaluate the effectiveness of the strategy. During the six months, CHWs will have weekly or bi-weekly contact with participants in-person or by phone to deliver the DECIDE modules and address social and economic needs.
  Arms: Patient Navigation+Diabetes Self-Management Support
Other: Standard Patient Navigation — Once the participant has completed the YCLS assessment with study staff, the navigator will receive the referral and follow-up with the participant to address the social and economic needs identified. The patient navigator will follow-up with the participant 2-3 times over the 6 months by phone or in-person about progress with the referral and help address additional needs that may develop during the 6-month intervention.
  Arms: Patient Navigation

SUMMARY:
In this pilot and feasibility study, the investigator will randomize 100 African-American, Hispanic, and/or Medicaid (all race/ethnicities) patients from KPNW with A1C ≥ 8 to one of two 6-month interventions: 1) patient navigation only; or 2) patient navigation + diabetes self-management training. Feasibility of a large-scale, pragmatic, randomized trial will be determined and preliminary effectiveness of treatment arms on A1C reduction among racial/ethnic minority and low-income patients with poorly managed diabetes will be examined.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to inform the design of a future large-scale, randomized trial that will test if there is added benefit to addressing both social and economic needs and diabetes self-management to improve diabetes management long-term among vulnerable populations. In this pilot, the investigator will randomize 100 African-American, Hispanic, and/or Medicaid (all race/ethnicities) patients from Kaiser Permanente Northwest (KPNW) with A1C ≥ 8 and poor follow-up in primary care to one of two 6-month interventions: 1) patient navigation only; or 2) patient navigation + diabetes self-management training. In both study arms, KPNW practice-embedded patient navigators will screen for medical, social and economic needs and connect participants to internal and external resources. In the second study arm, navigators will also refer participants to community health workers (CHWs) embedded in local community-based organizations, who will deliver diabetes self-management training. Feasibility of the full-scale trial will be based on several measures including recruitment, retention, success rate of referrals to navigators and CHWs, and whether medical, social, and/or economic needs are met. Qualitative interviews will be conducted with various stakeholders to assess intervention acceptability and determinants of implementation. Preliminary effects of A1C, diabetes-related care gaps, health care utilization, and medication adherence will also be examined. This pragmatic study design involves a collaborative effort among researchers, health system staff, health system senior leadership, and local community-based organizations. Findings from the full-scale trial will contribute critical knowledge on the most effective, sustainable model of care for integrating lay health workers in the efforts to improve diabetes management among high risk patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes diagnosis
* Current Kaiser Permanente Northwest member
* African-American, Hispanic/Latino (English, Spanish-speaking, or bilingual), and/or a Medicaid recipient (from any racial or ethnic background)
* Age 18 or older
* Most recent hemoglobin A1C test of ≥ 8
* Endorses 1 or more social and/or economic need on the Your Current Life Situation assessment

Exclusion Criteria:

* Patients who are unable to provide informed consent due to cognitive or psychiatric impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Fitzpatrick, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northwest, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papajorgji-Taylor D, Francisco M, Schneider JL, Vaughn K, Lindberg N, Smith N, Fitzpatrick SL. Bridge to Health/ Puente a la Salud: Rationale and design of a pilot feasibility randomized trial to address diabetes self-management and unmet basic needs among racial/ethnic minority and low-income patients. Contemp Clin Trials Commun. 2021 Apr 30;22:100779. doi: 10.1016/j.conctc.2021.100779. eCollection 2021 Jun. PMID 34013093
- [Result] Fitzpatrick SL, Papajorgji-Taylor D, Schneider JL, Lindberg N, Francisco M, Smith N, Vaughn K, Vrany EA, Hill-Briggs F. Bridge to Health/Puente a la Salud: a pilot randomized trial to address diabetes self-management and social needs among high-risk patients. Transl Behav Med. 2022 Jul 18;12(7):783-792. doi: 10.1093/tbm/ibac016. PMID 35849138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used a targeted recruitment approach by first identifying potentially eligible patients in the electronic health record (EHR) and then emailing or mailing recruitment letters. Letters were followed by a phone call from study staff who described the study and further assessed eligibility by confirming race/ethnicity and health coverage and administering a social risks screener.
Groups:
- Patient Navigation+Diabetes Self-Management Support: In addition to receiving navigation, participants in this arm will also be referred to Project Access NOW by study staff using REDCap. Project Access NOW will connect participants to a community-based organization based on their preference, previous experience with an agency, geography, and capacity.
  The CHW will follow-up with the participant to conduct a home visit and follow-up on community-based referrals already placed by the KPNW patient navigator and assess for additional needs. The timing of the diabetes self-management training will be based on the needs of the participant.
  Diabetes Self-Management Training: The Decision-making Education for Choices in Diabetes Everyday (DECIDE) program is a nine-module, literacy adapted diabetes and cardiovascular disease education and problem-solving training program. Participants are taught the five steps of problem solving with each module going in depth on a single step: 1) identify the problem; 2) brainstorm possible strategies for problem resolution; 3) select the most appropriate strategy; 4) apply the strategy; 5) evaluate the effectiveness of the strategy. During the six months, CHWs will have weekly or bi-weekly contract with participants in-person or by phone to deliver the DECIDE modules and address social and economic needs.
Period: Overall Study
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
Started | 54 | 56
Completed | 42 | 40
Not Completed | 12 | 16
Not completed — Lost to follow-up for intervention | 12 | 3
Not completed — Received only 1 component of intervention | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.1) | 53.7 (12.1) | 53.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 19 | 21 | 40
  Hispanic/Latino | 16 | 13 | 29
  Multiple Races | 1 | 2 | 3
  White | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 54 | 56 | 110
Primary Language [Count of Participants; unit: Participants]
  English | 46 | 50 | 96
  Spanish | 8 | 6 | 14
A1C [Mean (Standard Deviation); unit: % of glycosylated hemoglobin] | 9.9 (1.7) | 9.8 (1.6) | 9.9 (1.7)
Types of Social Needs Reported [Count of Participants; unit: Participants]
  Insufficient Housing | 15 | 18 | 33
  Financial Hardship | 51 | 45 | 96
  Food Insecurity | 34 | 33 | 67
  Lack of Transportation | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With A1C < 8%
Description: Using ITT analysis, percent of participants in each arm with A1C < 8% at 6-month follow-up was calculated.
Time Frame: 6 months
Population: ITT was used for primary outcome analysis so all participants included.
Measure: Number; unit: percent of participants
Groups:
- Patient Navigation+Diabetes Self-Management Support: In addition to receiving patient navigation, participants in this arm will also be referred to Project Access NOW by study staff using REDCap. Project Access NOW will connect participants to a community-based organization based on their preference, previous experience with an agency, geography, and capacity.
  The CHW will follow-up with the participant to conduct a home visit and follow-up on community-based referrals already placed by the KPNW patient navigator and assess for additional needs. The timing of the diabetes self-management training will be based on the needs of the participant.
  Diabetes Self-Management Training: The Decision-making Education for Choices in Diabetes Everyday (DECIDE) program is a nine-module, literacy adapted diabetes and cardiovascular disease education and problem-solving training program. Participants are taught the five steps of problem solving with each module going in depth on a single step: 1) identify the problem; 2) brainstorm possible strategies for problem resolution; 3) select the most appropriate strategy; 4) apply the strategy; 5) evaluate the effectiveness of the strategy. During the six months, CHWs will have weekly or bi-weekly contract with participants in-person or by phone to deliver the DECIDE modules and address social and economic needs.
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
Number analyzed (Participants) | 54 | 56
percent of participants | 33 | 34

2. Secondary Outcome: Emergency Department (ED) Visits
Description: Mean number of visits to the emergency department over the 6-month duration of the intervention.
Time Frame: 6 months
Population: Analysis for this secondary outcome includes all participants.
Measure: Mean (Standard Deviation); unit: visits
Groups:
- Patient Navigation+Diabetes Self-Management Support: In addition to receiving patient navigation, participants in this arm will also be referred to Project Access NOW by study staff using REDCap. Project Access NOW will connect participants to a community-based organization based on their preference, previous experience with an agency, geography, and capacity.The CHW will follow-up with the participant to conduct a home visit and follow-up on community-based referrals already placed by the KPNW patient navigator and assess for additional needs. The timing of the diabetes self-management training will be based on the needs of the participant.
  Diabetes Self-Management Training: The Decision-making Education for Choices in Diabetes Everyday (DECIDE) program is a nine-module, literacy adapted diabetes and cardiovascular disease education and problem-solving training program. Participants are taught the five steps of problem solving with each module going in depth on a single step: 1) identify the problem; 2) brainstorm possible strategies for problem resolution; 3) select the most appropriate strategy; 4) apply the strategy; 5) evaluate the effectiveness of the strategy. During the six months, CHWs will have weekly or bi-weekly contract with participants in-person or by phone to deliver the DECIDE modules and address social and economic needs.
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
Number analyzed (Participants) | 54 | 56
visits | 0.96 (1.70) | 1.07 (2.95)

3. Secondary Outcome: Primary Care Visit No-show Rate
Description: Mean number of missed primary care visits over duration of the intervention (6 months)
Time Frame: 6 months
Population: All participants were included in the analysis for this secondary outcome.
Measure: Mean (Standard Deviation); unit: missed visits
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
Number analyzed (Participants) | 54 | 56
missed visits | 0.85 (1.29) | 0.88 (1.62)

4. Secondary Outcome: Medication Refills
Description: Number of participants with 1 or more gaps in refilling oral diabetes medications during the study period. A gap is defined as not refilling prescription for 7 or more days after prescription has ran out.
Time Frame: 6 months
Population: Participants who were prescribed an oral diabetes medication during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
Number analyzed (Participants) | 45 | 45
Participants | 27 | 20

5. Secondary Outcome: Mean A1C Change
Description: Change in A1C from baseline to 6-month follow-up
Time Frame: 6 months
Population: ITT analysis was used for this outcome, so all participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
Number analyzed (Participants) | 54 | 56
percentage of glycosylated hemoglobin | 0.65 (1.76) | 0.72 (1.88)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 6 months for each participant; 2 years total for the overall study period.
Description: Adverse events were tracked using data from the electronic health record and based on the following events: hospitalizations, death, and hypoglycemia.
Arm/Group | Patient Navigation | Patient Navigation+Diabetes Self-Management Support
All-Cause Mortality (participants affected / at risk) | 1/54 | 1/56
Serious Adverse Events (participants affected / at risk) | 7/54 | 7/56
Other Adverse Events (participants affected / at risk) | 0/54 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Navigation (N=54) | Patient Navigation+Diabetes Self-Management Support (N=56)
Hospitalizations (Endocrine disorders) | 6 | 6 — If participants were hospitalized for any reasons related to having diabetes, then this was tracked as a serious adverse event.
Hypoglycemia (Endocrine disorders) | 1 | 1 — If a participant had a diagnosis of hypoglycemia (low blood sugar) for any medical encounter that occurred during the study period was considered a serious adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03802825/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03802825/SAP_001.pdf